CLINICAL TRIAL: NCT06586411
Title: Comparison of Oxygenation Index and Oxygen Stretch Index With Mechanical Power, Driving Pressure, Transpulmonary Pressure, and Lung Ultrasound Scores in PARDS Patients
Brief Title: Comparison of Oxygenation Index and Oxygen Stretch Index
Status: Completed | Type: Observational
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Collaborators: Hamilton Medical AG (Industry)
Responsible Party: Principal Investigator, Hasan ağın, Prof.Dr, Dr. Behcet Uz Children's Hospital
Other Study IDs: 02021/519
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Acute Respiratory Distress Syndrome
Keywords: Acute respiratory failure (ARF); Oxygenation index; Transpulmonary pressure; Mechanical power; Oxygen stretch index; Driving pressure; Lung ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PARDS: pediatric patients who were diagnosed with PARDS

SUMMARY:
Pediatric acute respiratory distress syndrome (pARDS) is a heterogeneous clinical syndrome that causes high rates of mortality and morbidity. The Pediatric Acute Lung Injury Consensus Conference (PALICC) guideline recommends using the oxygenation index (OI = mean airway pressure (MAP) × FiO2 /PaO2) for the diagnosis and classification of pediatric ARDS. Driving pressure (DP) is calculated by subtracting PEEP from plateau pressure. It is an important determinant of tidal volume in each breath and indirectly reflects lung stress.

It is the best parameter associated with mortality and lung injury in many studies. In the oxygenation index formula; adding driving pressure instead of Pmean may be more useful in evaluating the severity of pARDS. In our study, we will compare the Oxygenation Stress Index with OI in patients with pARDS. We will compare transpulmonary pressure, mechanical power, lung ultrasound score, and other respiratory mechanics, which are parameters indicating lung injury.

DETAILED DESCRIPTION:
Pediatric acute respiratory distress syndrome (pARDS) is a heterogeneous clinical syndrome that causes high rates of mortality and morbidity. The Pediatric Acute Lung Injury Consensus Conference (PALICC) guideline recommends using the oxygenation index (OI = mean airway pressure (MAP) × FiO2 /PaO2) for the diagnosis and classification of pediatric ARDS. In recent years, studies conducted on adult and pediatric populations have emphasized ''driving pressure'' as the most important ventilator parameter associated with mortality. Driving pressure (DP) is calculated by subtracting PEEP from plateau pressure. It is an important determinant of tidal volume in each breath and indirectly reflects lung stress. Lung stress is directly measured with transpulmonary pressure (PL).

Mechanical power (MP) is the amount of energy applied to patients per unit time and its relationship with lung injury has been shown in adult and pediatric studies. Another method that shows lung damage is measured noninvasively at the patient's bedside. It has been validated in many adult, pediatric, and neonatal studies. In an adult study, DP was used instead of MAP inspired by the oxygenation index and defined as the Oxygenation stretch index. It was emphasized that it can better predict oxygenation and mortality.

OI is not used in the ARDS classification in adults. Adding airway pressure to the oxygenation equation is very important to standardize the severity of the disease. However, its effect on patient outcomes has not been determined as much as mean airway pressure, plateau, and driving pressure. In addition, no target recommendation has been presented in the PALICC guidelines. Plateau pressure is the end-inspiratory pressure and does not have a direct effect on PEEP. Since ventilator management is still heterogeneous in pediatric literature in line with the guidelines, it seems more logical to use driving pressure, which includes both inspiratory pressure and expiratory pressure. Within the framework of this information, adding driving pressure to the formula instead of Pmean (MAP) in the oxygenation index may be useful in evaluating both the severity of pARDS and the effectiveness of respiratory dynamics.

In our study, we will compare the Oxygenation Stretch Index with OI in patients with pARDS. We will examine its effects on parameters indicating lung damage, respiratory mechanics and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* pARDS patient
* Intubated patient

Exclusion Criteria:

* Perinatal lung disease
* Cardiac failure and fluid overload
* Patients whose respiratory mechanics cannot be measured
* Age under 1 month or above 18 years old
* ETT leakage > 18%

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Intubated pARDS patients in PICU
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Correlation of Oxygenation Index and Oxygenation Stretch Index in Acute Pediatric Respiratory Distress Syndrome (pARDS) Patiens in the PICU | 2 hours
  By comparing the oxygenation stress index with the oxygenation index; it will be investigated whether it is a better parameter indicating lung damage. For this purpose, Oxygenation index and oxygenation stretch index will be correlated with mechanical power. Oxygenation index and oxygenation stretch index will be correlated with lung ultrasound score. Oxygenation index and oxygenation stretch index will be correlated with driving pressure. Oxygenation index and oxygenation stretch index will be correlated with transpulmonary pressure. Oxygenation index and oxygenation stretch index will be correlated with transpulmonary driving pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Agin, Study Chair — Dr. Behcet Uz Children's Hospital
Locations (6):
- Turkey (Türkiye) (6):
  - Aydin Obstetric and pediatrics Hospital, Aydin
  - Erzurum Regional Research and Training Hospital, Erzurum
  - Cam Sakura Research and Training Hospital, Istanbul
  - Acibadem University, Acibadem Altunizade Hospital, Istanbul
  - Istanbul Aydin University, Istanbul
  - The Health Sciences University Izmir Behçet Uz Child Health and Diseases Research and Training Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Schelven P, Koopman AA, Burgerhof JGM, Markhorst DG, Blokpoel RGT, Kneyber MCJ. Driving Pressure Is Associated With Outcome in Pediatric Acute Respiratory Failure. Pediatr Crit Care Med. 2022 Mar 1;23(3):e136-e144. doi: 10.1097/PCC.0000000000002848. PMID 34669679
- [Background] Emeriaud G, Lopez-Fernandez YM, Iyer NP, Bembea MM, Agulnik A, Barbaro RP, Baudin F, Bhalla A, Brunow de Carvalho W, Carroll CL, Cheifetz IM, Chisti MJ, Cruces P, Curley MAQ, Dahmer MK, Dalton HJ, Erickson SJ, Essouri S, Fernandez A, Flori HR, Grunwell JR, Jouvet P, Killien EY, Kneyber MCJ, Kudchadkar SR, Korang SK, Lee JH, Macrae DJ, Maddux A, Modesto I Alapont V, Morrow BM, Nadkarni VM, Napolitano N, Newth CJL, Pons-Odena M, Quasney MW, Rajapreyar P, Rambaud J, Randolph AG, Rimensberger P, Rowan CM, Sanchez-Pinto LN, Sapru A, Sauthier M, Shein SL, Smith LS, Steffen K, Takeuchi M, Thomas NJ, Tse SM, Valentine S, Ward S, Watson RS, Yehya N, Zimmerman JJ, Khemani RG; Second Pediatric Acute Lung Injury Consensus Conference (PALICC-2) Group on behalf of the Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Executive Summary of the Second International Guidelines for the Diagnosis and Management of Pediatric Acute Respiratory Distress Syndrome (PALICC-2). Pediatr Crit Care Med. 2023 Feb 1;24(2):143-168. doi: 10.1097/PCC.0000000000003147. Epub 2023 Jan 20. PMID 36661420
- [Background] Chen L, Chen GQ, Shore K, Shklar O, Martins C, Devenyi B, Lindsay P, McPhail H, Lanys A, Soliman I, Tuma M, Kim M, Porretta K, Greco P, Every H, Hayes C, Baker A, Friedrich JO, Brochard L. Implementing a bedside assessment of respiratory mechanics in patients with acute respiratory distress syndrome. Crit Care. 2017 Apr 4;21(1):84. doi: 10.1186/s13054-017-1671-8. PMID 28372575
- [Background] Chen L, Grieco DL, Beloncle F, Chen GQ, Tiribelli N, Madotto F, Fredes S, Lu C, Antonelli M, Mercat A, Slutsky AS, Zhou JX, Brochard L. Partition of respiratory mechanics in patients with acute respiratory distress syndrome and association with outcome: a multicentre clinical study. Intensive Care Med. 2022 Jul;48(7):888-898. doi: 10.1007/s00134-022-06724-y. Epub 2022 Jun 7. PMID 35670818
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Background] Khemani RG, Smith LS, Zimmerman JJ, Erickson S; Pediatric Acute Lung Injury Consensus Conference Group. Pediatric acute respiratory distress syndrome: definition, incidence, and epidemiology: proceedings from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5 Suppl 1):S23-40. doi: 10.1097/PCC.0000000000000432. PMID 26035358
- [Background] Mauri T, Yoshida T, Bellani G, Goligher EC, Carteaux G, Rittayamai N, Mojoli F, Chiumello D, Piquilloud L, Grasso S, Jubran A, Laghi F, Magder S, Pesenti A, Loring S, Gattinoni L, Talmor D, Blanch L, Amato M, Chen L, Brochard L, Mancebo J; PLeUral pressure working Group (PLUG-Acute Respiratory Failure section of the European Society of Intensive Care Medicine). Esophageal and transpulmonary pressure in the clinical setting: meaning, usefulness and perspectives. Intensive Care Med. 2016 Sep;42(9):1360-73. doi: 10.1007/s00134-016-4400-x. Epub 2016 Jun 22. PMID 27334266
- [Background] Chiumello D, Chidini G, Calderini E, Colombo A, Crimella F, Brioni M. Respiratory mechanics and lung stress/strain in children with acute respiratory distress syndrome. Ann Intensive Care. 2016 Dec;6(1):11. doi: 10.1186/s13613-016-0113-0. Epub 2016 Feb 5. PMID 26847436
- [Background] Vedrenne-Cloquet M, Khirani S, Khemani R, Lesage F, Oualha M, Renolleau S, Chiumello D, Demoule A, Fauroux B. Pleural and transpulmonary pressures to tailor protective ventilation in children. Thorax. 2023 Jan;78(1):97-105. doi: 10.1136/thorax-2021-218538. Epub 2022 Jul 8. PMID 35803726
- [Background] Khemani RG, Smith L, Lopez-Fernandez YM, Kwok J, Morzov R, Klein MJ, Yehya N, Willson D, Kneyber MCJ, Lillie J, Fernandez A, Newth CJL, Jouvet P, Thomas NJ; Pediatric Acute Respiratory Distress syndrome Incidence and Epidemiology (PARDIE) Investigators; Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Paediatric acute respiratory distress syndrome incidence and epidemiology (PARDIE): an international, observational study. Lancet Respir Med. 2019 Feb;7(2):115-128. doi: 10.1016/S2213-2600(18)30344-8. Epub 2018 Oct 22. PMID 30361119
- [Background] Mojoli F, Torriglia F, Orlando A, Bianchi I, Arisi E, Pozzi M. Technical aspects of bedside respiratory monitoring of transpulmonary pressure. Ann Transl Med. 2018 Oct;6(19):377. doi: 10.21037/atm.2018.08.37. PMID 30460251
- [Background] Ceylan G, Topal S, Atakul G, Colak M, Soydan E, Sandal O, Sari F, Agin H. Randomized crossover trial to compare driving pressures in a closed-loop and a conventional mechanical ventilation mode in pediatric patients. Pediatr Pulmonol. 2021 Sep;56(9):3035-3043. doi: 10.1002/ppul.25561. Epub 2021 Jul 22. PMID 34293255